CLINICAL TRIAL: NCT06926452
Title: Clinical and Volumetric Changes Following Single Pontic Site Development Using Multilayered Platelet Rich Fibrin Versus Connective Tissue Grafting in the Maxillary Esthetic Zone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Joseph Osama Joseph Kostandy, Post-graduate candidate in Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRF vs CTG
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Pontic Site Augmentation; Connective Tissue Graft
Keywords: Pontic site augmentation

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Procedure: Pontic site augmentation with sub-epithelial connective tissue graft.
- Test (Experimental)
  Interventions: Procedure: Pontic site augmenation using multi-layered platelet rich fibrin

INTERVENTIONS:
Procedure: Pontic site augmentation with sub-epithelial connective tissue graft. — Pontic site augmentation with sub-epithelial connective tissue graft.
  Arms: Control
Procedure: Pontic site augmenation using multi-layered platelet rich fibrin — Pontic site augmenation using multi-layered platelet rich fibrin
  Arms: Test

SUMMARY:
In clinical practice most patients' first concern is esthetics, soft tissue grafting is becoming routine in clinical practice to make up for the deficiency in supra-crestal tissue dimension that typically follows tooth loss. The edentulous site experiences major qualitative and quantitative changes because of a number of sequential events that occur after tooth extraction. Ridge dimensional alterations of the underlying bone and the soft tissue architecture overlaying it are the consequence of the socket healing process. To maintain the remaining teeth, aesthetic jaw support and optimal food chewing, lost teeth must be replaced. The teeth adjacent to and opposing a missing tooth will eventually tip, shift, and migrate, disrupting normal function. One integral part of the new strategy for treating periodontal diseases is thought to be surgical periodontal operations. Soft tissue grafting has become more frequently utilized to improve the aesthetics of teeth and dental implant sites by treating mucogingival abnormalities, restoring an appropriate width of keratinized tissue, and enhancing tissue thickness. SCTG has its own limitations, such as lack of graft availability, need for a second surgical site, proximity to palatine neurovascular complex and unaesthetic tissue contour at the recipient site. Due to these limitations, investigations on more regenerative nature techniques have been explored such as PRF, Using PRF instead of SCTG has the added value of decreasing discomfort and postoperative pain after the surgical procedure due to having additional donor site, To the best of our knowledge testing multi-layer PRF against SCTG in pontic site augmentation was never done before.

DETAILED DESCRIPTION:
In clinical practice most patients' first concern is esthetics, soft tissue grafting is becoming routine in clinical practice to make up for the deficiency in supra-crestal tissue dimension that typically follows tooth loss. The edentulous site experiences major qualitative and quantitative changes because of a number of sequential events that occur after tooth extraction. Ridge dimensional alterations of the underlying bone and the soft tissue architecture overlaying it are the consequence of the socket healing process. To maintain the remaining teeth, aesthetic jaw support and optimal food chewing, lost teeth must be replaced. The teeth adjacent to and opposing a missing tooth will eventually tip, shift, and migrate, disrupting normal function. One integral part of the new strategy for treating periodontal diseases is thought to be surgical periodontal operations. Soft tissue grafting has become more frequently utilized to improve the aesthetics of teeth and dental implant sites by treating mucogingival abnormalities, restoring an appropriate width of keratinized tissue, and enhancing tissue thickness. SCTG has its own limitations, such as lack of graft availability, need for a second surgical site, proximity to palatine neurovascular complex and unaesthetic tissue contour at the recipient site. Due to these limitations, investigations on more regenerative nature techniques have been explored such as PRF, Using PRF instead of SCTG has the added value of decreasing discomfort and postoperative pain after the surgical procedure due to having additional donor site, To the best of our knowledge testing multi-layer PRF against SCTG in pontic site augmentation was never done before.

Following tooth extraction, alveolar bone loss and structural and compositional changes of the covering soft tissues, as well as morphological alterations, can be expected. The numerous alterations in the alveolar process may lead to difficulties at the time of implant placement when a prosthetically driven implant position is desired, SCTG has its own limitations, such as lack of graft availability, need for a second surgical site, proximity to palatine neurovascular complex and unaesthetic tissue contour at the recipient site. The use of the SCTG in periodontal surgery is considered the golden pattern to the gingival recession treatment due to its characteristics of quick keratinization and adherence. However, the application of the technique is limited by the thickness of the giver tissue, anatomical factors, technical difficulty, and the need of an additional giver site. Due to these limitations, investigations on more regenerative nature techniques have been explored such as PRF. Platelet-Rich Fibrin (PRF) is an autologous biomaterial obtained from a patient's blood, rich in platelets, growth factors, and fibrin, which has regenerative and healing properties. Multi-layer PRF (ML-PRF) involves stacking several PRF membranes to increase their volumetric effect and improve tissue healing in areas requiring soft tissue augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Adults from the age of 18 - 40 years
* Patients with missing maxillary teeth/tooth in the area from 2nd premolar to 2nd premolar with ridge defect according to Seibert classification (Class I, II and III).
* Intact gingival tissue with at least 2mm keratinized tissue.
* Periodontally healthy patients.
* Patients accepts to provide informed consent.

Exclusion Criteria:

* Smokers.
* Pregnant females.
* Handicapped and mentally challenged patients.
* Systemic disease compromising wound healing.
* Active soft tissue infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Keratinized tissue thickness | 6 months

IPD SHARING:
Plan to Share IPD: Undecided